CLINICAL TRIAL: NCT00223951
Title: A Multi-Center, Randomized, Double-Masked, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety of R89674 0.25% Ophthalmic Solution in Healthy, Normal Volunteers
Brief Title: Safety Study of Ophthalmic Solution in Healthy, Normal Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vistakon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-003-10
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Volunteers Eligible for Study; Drug Being Developed for Allergic Conjunctivitis
Keywords: Healthy volunteers, safety, ocular, allergic conjunctivitis, ophthalmic
MeSH Terms: conditions — Conjunctivitis, Allergic

INTERVENTIONS:
Drug: R89674 (generic name not yet established)

SUMMARY:
The purpose of this study is to evaluate the safety of R89674 0.25% ophthalmic solution in healthy normal volunteers

ELIGIBILITY:
Inclusion Criteria:

healthy normal volunteers age >=3 years with normal ocular health and a best-corrected logMAR score of 0.3 or better

-

Exclusion Criteria:

intraocular surgery and/or ocular surgical intervention within last 3 months, refractive surgery within last 6 months, active ocular disorder other than refractive disorders, breastfeeding women, pregnant female < 18 years of age -

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900
Dates: Start 2005-09; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Adverse events; biomicroscopy and visual acuity at baseline and Days 7, 21, and 42; ophthalmoscopy and intraocular pressure at baseline and Day 42; physical examination

SECONDARY OUTCOMES:
No additional endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Jack V Greiner, OD, DO, PhD, Principal Investigator — Ophthalmic Research Associates, North Andover, MA
Locations (6):
- United States (6):
  - Phoenix, Arizona
  - Bel Air, Maryland
  - North Andover, Massachusetts
  - Las Vegas, Nevada
  - Charlotte, North Carolina
  - Philadelphia, Pennsylvania